CLINICAL TRIAL: NCT06228261
Title: Critical Analysis of the Results in the Management of Penetrating Abdominal Trauma in the Past Fifteen Years. Do we Need to Change the Protocol?
Brief Title: Critical Analysis of the Results in the Management of Penetrating Abdominal Trauma in the Past Fifteen Years.
Acronym: PAT-HMAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Doctor, Hospital del Mar
Other Study IDs: Penetrating abdotrauma HMAR
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Penetrating Abdominal Trauma
Keywords: Penetrating Trauma; Trauma surgery; Explorative laparoscopy; Trauma laparotomy; eFAST

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Penetrating abdominal trauma (PAT) incidence varies between 3,1-12,8% and it comprises a wide range of injuries with varying patterns on diagnostic imaging. Last guidelines published in 2014 recommend the use of FAST and CXR as the Gold Standard method for evaluating. Computed Tomography (CT) is widely used in stable patients with PAT and it requires intravenous contrast and patient irradiation, leading to additional costs to healthcare services. This study aims to assess the management of PAT in our institution and with its results review the actual protocol.

DETAILED DESCRIPTION:
Penetrating abdominal trauma (PAT) incidence varies between 3,1-12,8% and it comprises a wide range of injuries with varying patterns on diagnostic imaging. Last guidelines published in 2014 recommend the use of FAST and CXR as the Gold Standard method for evaluating. Computed Tomography (CT) is widely used in stable patients with PAT and it requires intravenous contrast and patient irradiation, leading to additional costs to healthcare services. This study aims to assess the management of PAT in our institution and with its results review the actual protocol.

A retrospective unicentric study will be conducted on a prospective database of stab wounds at the Department of General Surgery of Hospital del Mar over a 15-year period. The normality of the distribution of quantitative variables will be assessed using the Kolmogorov-Smirnov test. Comparison between qualitative variable groups will be performed using the Chi-square test or Fisher's exact test when appropriate, and non-parametric tests like the Mann-Whitney U test will be used to evaluate the significance of differences in means of quantitative variables. The odds ratios (OR) of predictor variables with outcome variables will be determined.

ELIGIBILITY:
Inclusion Criteria:

* All penetrating trauma patients admitted in the emergency department.

Exclusion Criteria:

* All patients with any other diagnostic different from penetrating trauma
* Blunt trauma patients admitted in the emergency department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a penetrating trauma in the neck admitted in Hospital del Mar from 2008 to 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Complications | 2008-2023
  The main outcome measure was the total of complications in patients with a penetrating abdominal trauma assessed by the Clavien-Dindo Classification.
Mortality | 2008-2023
  The second main outcome measure was the total of deaths in patients with a penetrating abdominal trauma assessed by preventable or non-preventable deaths.

SECONDARY OUTCOMES:
Explorations | 2008-2023
  To describe the explorations that has been ordered: eFAST, CT Scan, explorative laparoscopy or laparotomy.
Demographyc description | 2008-2023
  Description of the age and gender (Male / Female)
Physiologic description | 2008-2023
  Description of the vitals at arrival (bates per minute, blood pressure)
Wound and abdominal exploration | 2008-2023
  Description of the wound: bleeding, longitude, number of wounds and the abdominal explorations: peritonism or no peritonism.

CONTACTS AND LOCATIONS:
Overall Officials: Ana María González Castillo, PhD, Principal Investigator — Hospital del Mar

IPD SHARING:
Plan to Share IPD: No